CLINICAL TRIAL: NCT00373087
Title: Influence of Catechol-O-methyltransferase Polymorphism on Entacapone Efficacy in Parkinson's Disease
Brief Title: COMT Polymorphism and Entacapone Efficacy
Acronym: COMT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe Aucan, Department Clinical Research of Developpement
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P051034
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2007-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Catechol O-methyltransferase; Entacapone; pharmacogenetic
MeSH Terms: conditions — Parkinson Disease | interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-dopa + entacapone (Active Comparator): L-dopa + entacapone
  Interventions: Drug: entacapone
- L dopa / placebo (Experimental): L dopa / placebo
  Interventions: Drug: l dopa versus placebo

INTERVENTIONS:
Drug: entacapone — entacapone
  Arms: L-dopa + entacapone
Drug: l dopa versus placebo — l dopa versus placebo
  Arms: L dopa / placebo

SUMMARY:
Entacapone is an antiparkinsonian drug which block L-dopa metabolism, inhibiting the C-O-methyltransferase (COMT) enzyme. There is an individual variability of the COMT activity determined by a genetic polymorphism. The aim of this study is to investigate whether the genetic variability influences entacapone efficacy in Parkinson's disease.

DETAILED DESCRIPTION:
COMT protein is dependent of a single autosomal locus with two co-dominant alleles with a high activity (allele H) and a low activity (allele L) form of the enzyme. L and H allele frequency in the Caucasian population is around 50%. This is a monocentric randomized blinded cross-over study comparing acute challenge of L-dopa + placebo versus L-dopa + 200 mg entacapone, in Parkinson's disease patients with HH and LL genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* wearing off

Exclusion Criteria:

* atypical parkinsonism
* neuroleptic use

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
L-dopa efficacy duration on UPDRS motor scale during an acute L-dopa test | during the hospitalization in 24 hours
  L-dopa efficacy duration on UPDRS motor scale during an acute L-dopa test

SECONDARY OUTCOMES:
Pharmacokinetics of L-dopa and its metabolites | at the end of the study during the last hospitalization
  Pharmacokinetics of L-dopa and its metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe CORVOL, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Centre d'Investigation Clinique, Hôpital de la Pitié-Salpétrière,, Paris, France